CLINICAL TRIAL: NCT01846923
Title: Study of the B Memory Cell Response to Vaccination With the 13-valent Pneumococcal Conjugate Vaccine in Asplenic Individuals With Beta-thalassemia Major
Brief Title: B Memory Cell Response to Vaccination With the 13-valent Pneumococcal Conjugate Vaccine in Asplenic Individuals
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aghia Sophia Children's Hospital of Athens (Other)
Responsible Party: Principal Investigator, Vana Spoulou, Assistant Professor of Paediatrics, Aghia Sophia Children's Hospital of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 51657MoH
Record Dates: First submitted 2013-04-29; First posted 2013-05-06 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Asplenia; β-thalassemia Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PCV13 (Experimental)
  Interventions: Biological: PCV13

INTERVENTIONS:
Biological: PCV13

SUMMARY:
The purpose of this study is to determine whether one dose of the 13-valent pneumococcal conjugate vaccine (PCV13) induces immunological memory in asplenic adults and whether previously administered immunizations with the 23-valent polysaccharide pneumococcal vaccine influence the cellular immune response to PCV13 in this group.

ELIGIBILITY:
Inclusion Criteria:

* Asplenia
* β-thalassemia major
* older than 18 years

Exclusion Criteria:

* no previously recorded allergy to PCV
* no intravenous immunoglobulin (IVIG) given within the previous 6 months
* no other vaccine given within the previous 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2010-10; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
immunoglobulin G (IgG) B memory cell response one month post vaccination (measured by ELISpot) | One month post-PCV13
immunoglobulin M (IgM) B memory cell response one month post vaccination (measured by ELISpot) | one month post PCV13

SECONDARY OUTCOMES:
Maintenance of B memory cells three years after PCV13 vaccination | three years after study vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- 'Aghia Sophia' Children's Hospital, Athens, Attica, Greece

REFERENCES:
- [Derived] Papadatou I, Lagousi T, Kattamis A, Spoulou V. Antibody persistence 5 years after a 13-valent pneumococcal conjugate vaccine in asplenic patients with beta-thalassemia: assessing the need for booster. Ann Hematol. 2019 Mar;98(3):775-779. doi: 10.1007/s00277-019-03615-z. Epub 2019 Jan 25. PMID 30683996
- [Derived] Papadatou I, Piperi C, Alexandraki K, Kattamis A, Theodoridou M, Spoulou V. Antigen-specific B-cell response to 13-valent pneumococcal conjugate vaccine in asplenic individuals with beta-thalassemia previously immunized with 23-valent pneumococcal polysaccharide vaccine. Clin Infect Dis. 2014 Sep 15;59(6):862-5. doi: 10.1093/cid/ciu409. Epub 2014 May 30. PMID 24879786